CLINICAL TRIAL: NCT03029494
Title: The Role of Oxidative Stress and Opiorphin in Temporomandibular Disorders
Brief Title: Oxidative Stress and Opiorphin in Temporomandibular Disorders
Acronym: ROStrO-TMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Croatian Science Foundation (Other Government)
Responsible Party: Principal Investigator, Iva Alajbeg, Prof., University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IP- 2014-09-3070
Record Dates: First submitted 2017-01-19; First posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Temporomandibular Disorders
Keywords: oxidative stress; saliva
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Occlusal Splints; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: TMD patients will be randomized into two treatment groups. Each group will have two sets of interventions: one presumably active treatment and other a placebo:
  Treatment group 1: stabilization splint and placebo tablet daily. Treatment group 2: placebo (ineffectively designed) splint and 1000 mg Vitamin C tablet (an antioxidant agent) daily.
Who Masked: Participant
Masking Description: It will be a single-blind interventional study (as placebo splint cannot be mistaken for a stabilization splint by a clinician).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Treatment 1: stabilization splint, placebo oral tablet (Experimental): stabilization splint during night and 1 placebo oral tablet daily, for 6 months
  Interventions: Device: stabilization splint; Drug: Placebo Oral Tablet
- Treatment 2: placebo splint, vitamin C (Active Comparator): placebo splint during night and 1000 mg Vitamin C tablet daily, for 6 months
  Interventions: Device: placebo splint; Dietary Supplement: Vitamin C
- Control group (No Intervention): determination of oxidative stress biomarkers and cortisol in saliva of healthy control subjects

INTERVENTIONS:
Device: stabilization splint — Hard acrylic type of splint with full coverage of occlusal surfaces of upper teeth, with a thickness of about 1.5 mm at the level of the first molar.
  Other Names: occlusal splint
  Arms: Treatment 1: stabilization splint, placebo oral tablet
Drug: Placebo Oral Tablet — sugar pill manufactured to mimic 1000 mg Vitamin C
  Arms: Treatment 1: stabilization splint, placebo oral tablet
Device: placebo splint — Ineffectively designed oral appliance: an acrylic palatal plate will be used (without influence on occlusion, TMJ and masticatory muscles).
  Arms: Treatment 2: placebo splint, vitamin C
Dietary Supplement: Vitamin C — 1000 mg
  Other Names: ascorbic acid
  Arms: Treatment 2: placebo splint, vitamin C

SUMMARY:
The objective of this study is to quantify salivary oxidative stress biomarkers in patients with temporomandibular disorders and to quantify recently isolated endogenous peptide opiorphin in saliva of these patients. As chronic exposure to stress may cause hyperalgesia as a result of the stress response in the hypothalamic-pituitary-adrenal axis, aim is to test this as an underlying mechanism by correlating opiorphin and oxidative stress markers to salivary cortisol levels. The aim is to assess the association of oxidative stress salivary biomarkers with muscle and joint pain and to measure opiorphin, a potential biomarker of different pathological states.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) are most common chronic orofacial pain conditions of non-dental origin, with prevalence in the general population of 3.6% to 7%. Despite signs and symptoms being well described in the literature, there is still an absence of underlying pathophysiological mechanisms. Evidence based strategies for diagnosis and management of temporomandibular pain still aren't available. Psychological and mechanical stress factors could contribute to oxidative stress (OS) and lead to TMD. Therefore, identification of oxidative stress biomarkers would objectively indicate implication of OS in TMD pain onset mechanisms, and provide a basis for early detection, and a potential target for therapeutic agents to prevent progression to more severe dysfunction.

Aim is to quantify salivary OS markers and total antioxidant capacity (TAC), as well as recently isolated endogenous peptide opiorphin (OP) (2006 Inst. Pasteur), in TMD patients and compare them to controls. As chronic exposure to stress may cause hyperalgesia as a result of the stress response in the hypothalamic-pituitary-adrenal (HPA) axis, aim is to test this as an underlying mechanism by correlating OP and OS markers to salivary cortisol (SC) levels.

Hypotheses: OS has a role in TMD onset and maintenance, thus salivary markers of OS will increase and/or TAC will decrease; OP influences orofacial pain syndromes, such as TMD, and its salivary level will differ between TMD patients and controls. If decreased OP levels in TMD patients were encountered, we hypothesize that OP downregulation contributes to TMD onset as its analgesic effect is absent. Conversely, increased OP levels would suggest that OP is upregulated merely as a reaction to painful stimuli. Disbalanced SC levels in TMD patients would corroborate involvement of HPA axis in TMD mechanism, which is known to affect the intensity of OS.

Saliva of 50 TMD patients (diagnosed by validated diagnostic criteria and MRI) and 50 controls will be collected. OS markers (8-hydroxydeoxyguanosine, malondialdehyde, etc.) will be assessed by ELISA with spectrophotometric detection and by spectrophotometric reagent kits. OP levels will be measured by HPLC-MS/MS method, originally developed and validated by team members. The electrochemiluminescence immunoassay ECLIA will be used for measuring SC.

Pain and stress will be subjectively assessed using questionnaires: all subjects will fill in Perceived Stress Scale 10 (PSS-10); in TMD patients the worst experienced pain will be recorded using Visual Analogue Scale at the initial and at subsequent visits, as well as Graded Chronic Pain Scale (GCPS), Visual Analogue Scale (VAS), Patient Health Questionnaire (PHQ), Jaw function limitation scale (JFLS), Oral Behaviours Checklist and Oral Health Impact Profile (OHIP)-14.

TMD patients will be randomized in 2 treatment groups (1: stabilization splint + placebo pills; 2: placebo splint + 1g of vitamin C daily). Measurements will be repeated after 3 and 6 months of treatment. Monitoring of OP, OS markers and SC during that period will, depending on observed changes in TMD symptoms, further elucidate underlying proposed mechanism by performing multivariate analyses including treatment outcomes.

This translational research aims to make basic science findings useful for clinical applications. Findings of higher concentrations of OS biomarkers would, besides their significance as "a piece of puzzle" of TMD mechanism, could also be important in establishment of TMD diagnosis and as prospective therapeutic targets. Salivary opiorphin, due to its proven analgesic effect might additionally serve as a possible drug for orofacial pain syndromes.

Novel approach to understanding neuroendocrine mechanisms in TMD and their links to OS, as well and use of saliva as non-invasively available diagnostic biofluid represent significant scientific advances.

ELIGIBILITY:
Inclusion Criteria:

* for TMD patients: diagnosis of TMD using Croatian version of research diagnostic criteria for temporomandibular disorders (RDC/TMD)
* for control group: gender- and age-matched healthy volunteers

Exclusion Criteria:

* for TMD patients: patients younger than 18 years; smoking; other local diseases and/or systemic disorders; the use of anti-inflammatory drugs, analgesics and/or muscle relaxants; individuals who had already been under treatment for TMD
* for control group: younger than 18 years; cardiac/circulatory/metabolic/muscle abnormalities; smoking; the use of medications, supplements or dietary aids that might affect the outcome results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of salivary oxidative stress markers concentration | baseline, 6th month
  Oxidative stress markers will be measured using spectrophotometric methods. Opiorphin levels will be measured by HPLC-MS/MS method, originally developed and validated by team members (Brkljacic L, Sabalic M, Salaric I, Jeric I, Alajbeg I et al, J Chromatogr B Analyt Technol Biomed Life Sci. 2011). The change of the single marker (opiorphin) concentration between the two time points is a measure of clinical efficacy of applied treatment modality.
  In control group (healthy patients) measurement of oxidative stress markers and opiorphin will be performed only at first appointment in order to compare them with TMD patients baseline levels.

SECONDARY OUTCOMES:
Change of pain intensity in TMD patients | baseline, 3rd month, 6th month
  The intensity of pain will be determined using a 100 mm visual analog scale (VAS) on day 0, day 90 and day 180. The change in the amount between the time points is a measure of clinical efficacy of applied treatment modality.
The quality of life change in TMD patients | baseline, 6th month
  The quality of life for OLP patients will be determined using "Oral health impact profile"(OHIP-14) questionnaire on day 0 and day 180. The change in the amount between the time points is a measure of clinical efficacy of applied treatment modality.
Change in the amount of maximal comfortable mouth opening in TMD patients | baseline, 6th month
  Maximal comfortable mouth opening is measured as the distance between the maxillary and mandibular incisal edges. Maximal comfortable opening is defined as the maximum distance the participant could open his/her mouth without experiencing any additional pain and discomfort. The change in the amount of maximal comfortable mouth opening between the time points is a measure of clinical efficacy of applied treatment modality.
Change in the perceived stress | baseline, 6th month
  General anxiety disorder (GAD - 7) scale will be used in order to determine how often the patient has been disturbed by different problems including feeling of nervousness and anxiety. The change in the amount between the time points is a measure of clinical efficacy of applied treatment modality. In control group (healthy patients) GAD-7 will be used only at first appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Iva Z Alajbeg, PhD, Principal Investigator — School of Dental Medicine, University of Zagreb
Locations (1):
- School of Dental Medicine, University of Zagreb, Zagreb, N/A = Not Applicable, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] De Leeuw R, Bertoli E, Schmidt JE, Carlson CR. Prevalence of post-traumatic stress disorder symptoms in orofacial pain patients. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 May;99(5):558-68. doi: 10.1016/j.tripleo.2004.05.016. PMID 15829878
- [Result] De Leeuw R, Bertoli E, Schmidt JE, Carlson CR. Prevalence of traumatic stressors in patients with temporomandibular disorders. J Oral Maxillofac Surg. 2005 Jan;63(1):42-50. doi: 10.1016/j.joms.2004.04.027. PMID 15635556
- [Result] Kawai Y, Kubota E, Okabe E. Reactive oxygen species participation in experimentally induced arthritis of the temporomandibular joint in rats. J Dent Res. 2000 Jul;79(7):1489-95. doi: 10.1177/00220345000790071001. PMID 11005733
- [Result] Rodriguez de Sotillo D, Velly AM, Hadley M, Fricton JR. Evidence of oxidative stress in temporomandibular disorders: a pilot study. J Oral Rehabil. 2011 Oct;38(10):722-8. doi: 10.1111/j.1365-2842.2011.02216.x. Epub 2011 Apr 4. PMID 21457291
- [Result] Salaric I, Sabalic M, Alajbeg I. Opiorphin in burning mouth syndrome patients: a case-control study. Clin Oral Investig. 2017 Sep;21(7):2363-2370. doi: 10.1007/s00784-016-2031-9. Epub 2016 Dec 24. PMID 28013436
- [Result] Turp JC, Komine F, Hugger A. Efficacy of stabilization splints for the management of patients with masticatory muscle pain: a qualitative systematic review. Clin Oral Investig. 2004 Dec;8(4):179-95. doi: 10.1007/s00784-004-0265-4. Epub 2004 Jun 4. PMID 15179561
- [Result] Miricescu D, Totan A, Calenic B, Mocanu B, Didilescu A, Mohora M, Spinu T, Greabu M. Salivary biomarkers: relationship between oxidative stress and alveolar bone loss in chronic periodontitis. Acta Odontol Scand. 2014 Jan;72(1):42-7. doi: 10.3109/00016357.2013.795659. Epub 2013 Jul 22. PMID 23869629
- [Result] Lawaf S, Azizi A, Tabarestani T. Comparison of Serum and Salivary Antioxidants in Patients with Temporomandibular Joint Disorders and Healthy Subjects. J Dent (Tehran). 2015 Apr;12(4):263-70. PMID 26622281
- [Result] Wang J, Schipper HM, Velly AM, Mohit S, Gornitsky M. Salivary biomarkers of oxidative stress: A critical review. Free Radic Biol Med. 2015 Aug;85:95-104. doi: 10.1016/j.freeradbiomed.2015.04.005. Epub 2015 Apr 16. PMID 25889823
- [Derived] Vrbanovic E, Lapic I, Rogic D, Alajbeg IZ. Changes in salivary oxidative status, salivary cortisol, and clinical symptoms in female patients with temporomandibular disorders during occlusal splint therapy: a 3-month follow up. BMC Oral Health. 2019 Jun 6;19(1):100. doi: 10.1186/s12903-019-0791-8. PMID 31170954
- [Derived] Alajbeg IZ, Lapic I, Rogic D, Vuletic L, Andabak Rogulj A, Illes D, Knezovic Zlataric D, Badel T, Vrbanovic E, Alajbeg I. Within-Subject Reliability and between-Subject Variability of Oxidative Stress Markers in Saliva of Healthy Subjects: A Longitudinal Pilot Study. Dis Markers. 2017;2017:2697464. doi: 10.1155/2017/2697464. Epub 2017 Nov 15. PMID 29269980